CLINICAL TRIAL: NCT02758275
Title: Efficacy of Nursing Intervention "Teaching: Individual" to Increase Adherence to Therapeutic Regimen in People With Hypertension Arterial and/or Diabetes Mellitus Type 2
Brief Title: Teaching: Individual to Increase Adherence to Therapeutic Regimen in Hypertension Arterial and/or Diabetes Type 2
Acronym: ENURSIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Industrial de Santander (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); Cardiecol (Unknown); Instituto de Salud de Bucaramanga (Other)
Responsible Party: Principal Investigator, Sandra Lucrecia Romero Guevara, Nurse Research, MSc Nursing. Professor, School of Nursing. Universidad Industrial de Santander, Bucaramanga, Colombia., Universidad Industrial de Santander
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1861
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: Medication adherence; Patient compliance; Diabetes mellitus, Type 2; Hypertension; Nursing; Nursing process; Teaching; Randomized controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Medication Adherence; Patient Compliance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teaching: Individual (5606) (Experimental): People will receive an education session per month for a period of six months with an average duration of 30 minutes. These will be performed by nurses outside the collection of phase base line and follow-up measurements, previously trained for the purpose.
  Interventions: Behavioral: Teaching: Individual (5606)
- Usual care (No Intervention): People will continue to receive usual care in the health center where they usually assist to medical controls.

INTERVENTIONS:
Behavioral: Teaching: Individual (5606) — Usual care and Teaching: Individual (5606): It consists of 6 educational sessions:
  1. Behavior Modification (4360) Promotion of a behavior change.
  2. Teaching Disease Process (5602) Assisting the patient to understand information related to a specific disease process.
  3. Teaching: Prescribed Medication (5616) Preparing a patient to safely take prescribed medications and monitor for their effects.
  4. Teaching: Prescribed Diet (5614) Preparing a patient to correctly follow a prescribed diet.
  5. Teaching: Prescribed Exercise (5612) Preparing a patient to achieve and/or maintain a prescribed level of activity.
  6. Coping Enhancement (5230) Assisting a patient to adapt to perceived stressors, changes, or threats that interfere with meeting life demands and roles.
  Arms: Teaching: Individual (5606)

SUMMARY:
The purpose of this study is to improve the adherence of therapeutic regimen in people with hypertension arterial and/or diabetes mellitus type 2. Our hypothesis is the nursing intervention "Teaching: Individual", is more effective to increase adherence of therapeutic regimen in people with hypertension arterial and/or diabetes mellitus type 2, than usual care.

DETAILED DESCRIPTION:
Introduction: The hypertension arterial and diabetes mellitus are chronic diseases with a high burden of disease. It affects approximately 25% of the adult population worldwide and is an important risk factors for global mortality. As for the diabetes, worldwide there are about 346 million people with diabetes and 80% of them live in countries with low and middle income. The recommendations for treating of these diseases includes the pharmacological treatment and modification of lifestyle: salt restriction, moderation in alcohol consumption, high consumption of fruits and vegetables, low-fat diet, weight reduction and regular physical activity. The adherence to these guidelines are essential keys to success in handling these pathologies. The lack of adherence to the prescribed treatment regimen remains a problem among patients with long-term treatment.

Objective: To evaluated the efficacy of nursing intervention "Teaching: Individual" compared with usual care, to increase adherence of therapeutic regimen in people with hypertension arterial and/or diabetes mellitus type 2.

Methods: Randomized controlled trial. 200 patients with hypertension arterial and/or diabetes mellitus type 2 attending cardiovascular risk programs of Bucaramanga, Colombia will include . Nursing intervention to evaluate is "Teaching: Individual" consisting in six educational sessions. The investigators will measure 0, 6 y 12 months: Treatment Behavior: Illness or Injury (1609) (adherence treatment), glycosylated hemoglobin (HbA1c) and systolic blood pressure for 24 hours. Base characteristics of the groups will be compare through chi-square/Fisher´s exact or Students-T/Mann-Whitney U test. Outcomes will be evaluate by paired T-tests or Wilcoxon test at different follow-up times and statistical significance with p-value < 0.05 will considered.

ELIGIBILITY:
Inclusion Criteria:

* Adult population ≥ 18 years old
* Medical diagnosis of hypertension arterial and/or diabetes mellitus type 2.
* Attendees cardiovascular risk programs of Empresa Social del Estado Instituto de Salud de Bucaramanga (ISABU)
* People totally independent of their care.
* Access to a fixed telephone line or mobile itself
* Be residents of Bucaramanga

Exclusion Criteria:

* Changes in the mental sphere. Abbreviated Mental Test (Minimental) and Yesavage depression test.
* Communication limitations or chronic or serious alterations that make it hard compression of interventions.
* Subjects who are participating in a research study currently or during the last six months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Changes of mean score adherence to treatment from baseline at 6 and 12 months | 6 and 12 months
  Measured by Treatment Behavior: Illness or Injury (1609)

SECONDARY OUTCOMES:
Changes of mean score glycosylated hemoglobin from baseline at 6 and 12 months | 6 and 12 months
  Measured in peripheral venous blood
Changes of mean systolic blood pressure from baseline at 6 and 12 months | 6 and 12 months
  Measured by ambulatory blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Lucrecia SL Romero Guevara, MSc Nursing, Principal Investigator — Universidad Industrial de Santander; Dora Inés DI Parra, MSc Nursing, Principal Investigator — Universidad Industrial de Santander
Locations (2):
- Colombia (2):
  - Empresa Social del Estado Instituto de Salud de Bucaramanga (ESE ISABU), Bucaramanga, Santander Department
  - Nursing School, Universidad Industrial de Santander, Bucaramanga, Santander Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Romero S, Parra D, Sánchez J, Rojas L. Adherence to therapeutic regimen of hypertension andtype-2 diabetes patients in Bucaramanga, Colombia . Rev Univ Ind Santander Salud. 2017; 49(1): 37-44. DOI: http://dx.doi.org/10.18273/revsal.v49n1-2017004
- [Result] López L, Romero S, Parra D, Rojas L. Adherence to treatment: concept and measurement. Hacia promoc. salud. 2016; 21(1): 117-137. DOI: 10.17151/hpsal.2016.21.1.10
- [Derived] Romero Guevara SL, Parra DI, Rojas LZ. "Teaching: Individual" to increase adherence to therapeutic regimen in people with hypertension and type-2 diabetes: protocol of the controlled clinical trial ENURSIN. BMC Nurs. 2019 Jun 4;18:22. doi: 10.1186/s12912-019-0344-0. eCollection 2019. PMID 31171916